CLINICAL TRIAL: NCT05046353
Title: D-serine Augmentation of Neuroplasticity-based Auditory Learning in Schizophrenia: R33 Phase
Brief Title: D-serine AudRem: R33 Phase
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: U.S. Department of Health and Human Services OHRP issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023. NKI site is open for enrollment.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Nathan Kline Institute for Psychiatric Research (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joshua Kantrowitz, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7725R
Record Dates: First submitted 2021-08-30; First posted 2021-09-16 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia; Schizo Affective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- D-serine (Experimental): Subjects will receive 16 sessions of auditory remediation paired with either D-serine or Placebo in a 1:1 D-serine 120 mg/kg:placebo ratio.
  Interventions: Drug: D-serine
- placebo (Placebo Comparator): Subjects will receive 16 sessions of auditory remediation paired with either D-serine or Placebo in a 1:1 D-serine 120 mg/kg:placebo ratio.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: D-serine — Auditory remediation +/-D-serine
  Arms: D-serine
Other: Placebo — Auditory remediation +/-D-serine
  Arms: placebo

SUMMARY:
Schizophrenia is a major public health problem associated with cognitive deficits, such as short and long term memory, executive functioning, attention and speed of processing that are amongst the strongest predictors of impaired functional outcome. In addition, schizophrenia patients show reduced "plasticity", defined as reduced learning.

D-serine is a naturally occurring activator of the N-methyl-d-aspartate-type glutamate receptors (NMDAR) in the brain, and this project will assess the D-serine treatment over 16 weeks of a program designed to measure auditory plasticity.

DETAILED DESCRIPTION:
D-Serine is a naturally occurring substance in the brain that activates the N-methyl-d-aspartate-type glutamate receptor (NMDAR). This receptor is thought to be important in both schizophrenia and plasticity (learning). My model proposes that problems with NMDAR within the brain leads to impaired plasticity, which in turn leads to impaired cognition. d-serine is an ideal NMDAR activator to study because it balances efficacy, availability and safety. Most d-serine studies have used a low dose, but the evidence for efficacy is even stronger for high dose d-serine, as will be tested in the current study. There has only been limited summary of higher dose d-serine, which is another important reason for this study.

In addition to testing a potentially viable treatment in schizophrenia, a positive result would provide opportunities for use of D-serine in other populations (e.g. anxiety disorders or dementia) and stimulate the pharmaceutical industry to utilize this methodology to assess the efficacy of novel NMDAR modulators, using d-serine as a "gold-standard."

The ultimate goal of this two part grant (R61-R33) study is to improve cognitive remediation by augmenting with D-serine.

We recently completed the R61-phase, meeting our predetermined "milestones. " As predicted, D-serine led to significant enhancement of auditory plasticity and electrophysiological measures.

During the three-year R33-phase, we will conduct a study of D-serine of 60 schizophrenia patients, assessing the effects of D-serine over 16 sessions of this program. Most successful, cognitive remediation programs are limited by lengthy (30-50 hours) treatments. Hypothesizing that adding D-serine will increase efficiency of cognitive remediation, successful completion of the R33-phase is defined as significant improvement in global cognition after 16 hours of treatment, and will serve as a pilot study to determine whether future, definitive clinical trials are warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50
2. DSM-V diagnosis of schizophrenia or schizoaffective disorder
3. Willing to provide informed consent
4. Auditory Cognitive impairment demonstrated by:

   a .MCCB composite domain score less than or equal to 0.5 standard deviation below normal (T score less than or equal to 45) b. And at least one of the following:
5. MCCB verbal memory domain score less than or equal to 0.5 standard deviation below normal (T score less than or equal to 45)
6. Tone matching score of less than or equal to 77.7%
7. Clinically stable for 2 months (CGI less than or equal to 4)
8. Moderate or lower cognitive disorganization (PANSS P2 less than or equal to 4)
9. Medically stable for study participation
10. Willing to use qualified methods of contraception for the study duration and up to 2 months after its end
11. Fluent English speaker
12. Normal hearing
13. Visual acuity corrected to 20/30
14. An estimated Glomerular Filtration Rate (GFR) greater than or equal to 60
15. Taking an antipsychotic medication other than clozapine at a stable dose for at least 4 weeks
16. Judged clinically not to be at significant suicide or violence risk

Exclusion Criteria:

1. Substance abuse (excluding nicotine) within last 60 days
2. ECG abnormality that is clinically significant in the context of study participation in the opinion of the study cardiologist
3. Current clozapine use. Clozapine is excluded for two reasons: to avoid the potential confound of treatment resistant patients and because of clozapine's intrinsic NMDA agonist
4. Participation in study of investigational medication/device within 4 weeks
5. Pregnant women or women of child-bearing potential, who are either not surgically-sterile or for outpatients, using appropriate methods of birth control. Women of child-bearing potential must have a negative serum beta-hCG pregnancy test at screening.
6. Presence of positive history of unstable significant medical or neurological illness
7. Positive toxicology screen for any substances of abuse
8. Subjects with suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the Suicidal Ideation section of the baseline C-SSRS) in the 6 months prior to screening or subjects who represent a significant risk of suicide in the opinion of the investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Auditory Cognition | 16 weeks
  MATRICS cognitive battery verbal domain

CONTACTS AND LOCATIONS:
Locations (1):
- NYSPI, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will likely be available at https://nda.nih.gov